CLINICAL TRIAL: NCT06130540
Title: An Open-label, Multicenter Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Intravenous Secukinumab Infusion in Adults With Giant Cell Arteritis (GCA) or Polymyalgia Rheumatica (PMR)
Brief Title: Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Intravenous Secukinumab in Patients With GCA or PMR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457E22101; 2023-507667-19-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Giant Cell Arteritis; Polymyalgia Rheumatica
Keywords: Giant cell arteritis (GCA); Polymyalgia rheumatica (PMR); Secukinumab; pharmacokinetics; intravenous
MeSH Terms: conditions — Giant Cell Arteritis; Polymyalgia Rheumatica | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: 30 patients per cohort (Giant Cell Arteritis (GCA) and Polymyalgia Rheumatica (PRM) are planned to be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab: Giant Cell Arteritis (GCA) (Experimental)
  Interventions: Drug: Secukinumab
- Secukinumab: Polymyalgia Rheumatica (PMR) (Experimental)
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Intravenous (i.v.) doses of Secukinumab at Week 0, Week 4 and Week 8
  Other Names: AIN457

SUMMARY:
This study will examine how intravenous (i.v.) Secukinumab will be processed in the body (pharmacokinetics [PK]) and whether it will be safe and tolerable after multiple doses of i.v. Secukinumab infusion in adult patients with giant cell arteritis (GCA) or polymyalgia rheumatica (PMR).

DETAILED DESCRIPTION:
This is a 12-week, open-label, multicenter, basket design study followed by an 8-week follow-up period in two cohorts of participants, one cohort with GCA and one cohort with PMR.

This study will consist of 3 phases: screening, treatment and follow-up.

Participants will enter a screening period: up to 6 weeks to assess eligibility [or up to 8 weeks in the event of a major healthcare disruption or a need to complete screening requirements (e.g., required washouts, TB testing, and work up and treatment as needed per local guidelines. Participants will enter a treatment period of 12 weeks: 2 cohorts (GCA and PMR cohorts) receiving total of 3 i.v. doses of Secukinumab (Week 0, Week 4 and Week 8). After treatment participants will enter a follow-up period: 8 weeks treatment-free follow-up (12 weeks after last dose of study treatment).

The total duration of the trial for a participant (from screening to follow up) is approximately 26 weeks (maximum of approximately 28 weeks) including safety follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

Inclusion Criteria for GCA:

1. Male or non-pregnant, non-lactating female participants at least 50 years of age
2. Diagnosis of GCA based on meeting all of the following criteria:

   * Unequivocal cranial symptoms of GCA (e.g., new-onset localized headache, scalp or temporal artery tenderness, permanent or temporary ischemia-related vision loss, or otherwise unexplained mouth or jaw pain upon mastication), and/or unequivocal symptoms of PMR (defined as shoulder and/or hip girdle pain associated with inflammatory morning stiffness) and/or symptoms of limb ischemia (claudication)
   * Temporal artery biopsy (TAB) revealing features of GCA and/or cross-sectional imaging study such as ultrasound (e.g., cranial or axillary), MRI/MRA, CTA, or PET-CT with evidence of vasculitis
3. Active GCA disease within 6 months prior to Baseline as defined by meeting both of the following:

   * Presence of signs or symptoms attributed to active GCA and not related to prior damage (e.g., vision loss that occurred without new findings)
   * Elevated ESR >= 30 mm/hr or CRP >= 10 mg/L attributed to active GCA or active GCA on TAB or on imaging study

Inclusion Criteria for PMR:

1. Male or non-pregnant, non-lactating female participants at least 50 years of age
2. Diagnosis of PMR according to the provisional ACR/EULAR classification criteria: Participants >= 50 years of age with a history of bilateral shoulder pain accompanied by elevated CRP concentration (>= 10 mg/L) and/or elevated ESR (>= 30 mm/hr) who scored at least 4 points from the following optional classification criteria:

   * Morning stiffness >45 min (2 points)
   * Hip pain or restricted range of motion (1 point)
   * Absence of rheumatoid factor and/or anti-citrullinated protein antibodies (2 points)
   * Absence of other joint involvement (1 point)
3. Active PMR disease within 6 months prior to Baseline as defined by signs and symptoms attributable to PMR meeting the following:

   * Bilateral shoulder girdle and/or bilateral hip girdle pain associated with inflammatory stiffness with or without additional symptoms indicative of a PMR relapse (such as constitutional symptoms) that are in the opinion of the Investigator not due to other diseases that may mimic PMR such as osteoarthritis in shoulders or hips, polyarticular calcium pyrophosphate deposition disease, rotator cuff disease, adhesive capsulitis (frozen shoulder) or fibromyalgia

Key Exclusion Criteria:

Exclusion Criteria for GCA:

1. Pregnant or nursing (lactating) women where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
2. History of hypersensitivity or contraindication to any of the study treatments or its excipients or to drugs of similar chemical classes
3. Use of other investigational drugs within 5 half-lives of enrollment or within 30 days (e.g., small molecules) or until the expected pharmacodynamic effect has returned to BSL (e.g., biologics), whichever is longer; or longer if required by local regulations
4. History of clinically significant liver disease or liver injury as indicated by clinically significantly abnormal liver function tests (LFTs), such as SGOT (AST), SGPT (ALT) and serum bilirubin. The Investigator should be guided by the following criteria:

   * AST (Aspartate Aminotransferase) and ALT (Alanine Aminotransferase) may not exceed 3 x the upper limit of normal (ULN)
   * Total bilirubin concentration may not exceed 1.5 x ULN Any one of these parameters, if elevated above ULN, should be re-checked once more as soon as possible, and in all cases, at least prior to enrollment, to rule-out laboratory error.
5. Active infections or history of ongoing, chronic or recurrent infectious disease including but not limited to below:

   * Active infections during the last 2 weeks prior to BSL
   * Known infection with human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV) at screening or BSL, except for HCV successfully treated and cured, according to local/global guidelines
   * Evidence of tuberculosis (TB) infection as defined by a positive QuantiFERON TB-Gold Plus test. Participants with a positive test may participate in the study if further work-up (according to local practice/guidelines) establishes conclusively that the participant has no evidence of active TB. If the test result is indeterminate, the Investigator may repeat the test once or may proceed directly to perform the work-up for TB as per local procedures. If presence of latent TB is established, then treatment must be initiated prior to BSL (both treatment and timing prior to BSL according to local country guidelines)
6. Active inflammatory bowel disease or active uveitis
7. Active ongoing diseases which in the opinion of the Investigator immuno-compromises the participant and/or places the participant at unacceptable risk for treatment with immunomodulatory therapy
8. Current severe progressive or uncontrolled disease, which in the judgment of the Investigator renders the participant unsuitable for the trial, including but not limited to below:

   * Major ischemic event (e.g., myocardial infarction, stroke, etc.) or transient ischemic attack (TIA) within 12 weeks of screening
   * Significant medical conditions or diseases, including but not limited to the following: uncontrolled hypertension, congestive heart failure (New York Heart Association (NYHA) status of class III or IV) and uncontrolled diabetes mellitus
   * Any other current severe progressive or uncontrolled diseases per the Investigator's discretion
9. Confirmed diagnosis of any primary form of systemic vasculitis, other than GCA

Exclusion Criteria for PMR:

1. Pregnant or nursing (lactating) women where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
2. History of hypersensitivity or contraindication to any of the study treatments or its excipients or to drugs of similar chemical classes
3. Use of other investigational drugs within 5 half-lives of enrollment or within 30 days (e.g., small molecules) or until the expected pharmacodynamic effect has returned to BSL (e.g., biologics), whichever is longer; or longer if required by local regulations
4. History of clinically significant liver disease or liver injury as indicated by clinically significantly abnormal liver function tests (LFTs), such as SGOT (AST), SGPT (ALT) and serum bilirubin. The Investigator should be guided by the following criteria:

   * AST (Aspartate Aminotransferase) and ALT (Alanine Aminotransferase) may not exceed 3 x the upper limit of normal (ULN)
   * Total bilirubin concentration may not exceed 1.5 x ULN Any one of these parameters, if elevated above ULN, should be re-checked once more as soon as possible, and in all cases, at least prior to enrollment, to rule-out laboratory error.
5. Active infections or history of ongoing, chronic or recurrent infectious disease including but not limited to below:

   * Active infections during the last 2 weeks prior to BSL
   * Known infection with human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV) at screening or BSL, except for HCV successfully treated and cured, according to local/global guidelines
   * Evidence of TB infection as defined by a positive QuantiFERON TB-Gold Plus test. Participants with a positive test may participate in the study if further work-up (according to local practice/guidelines) establishes conclusively that the participant has no evidence of active TB. If the test result is indeterminate, the Investigator may repeat the test once or may proceed directly to perform the work-up for TB as per local procedures. If presence of latent TB is established, then treatment must be initiated prior to BSL (both treatment and timing prior to BSL according to local country guidelines)
6. Active inflammatory bowel disease or active uveitis
7. Active ongoing diseases which in the opinion of the Investigator immuno-compromises the participant and/or places the participant at unacceptable risk for treatment with immunomodulatory therapy
8. Current severe progressive or uncontrolled disease, which in the judgment of the Investigator renders the participant unsuitable for the trial, including but not limited to below:

   * Major ischemic event (e.g., myocardial infarction, stroke, etc.) or transient ischemic attack (TIA) within 12 weeks of screening
   * Significant medical conditions or diseases, including but not limited to the following: uncontrolled hypertension, congestive heart failure (New York Heart Association (NYHA) status of class III or IV) and uncontrolled diabetes mellitus
   * Any other current severe progressive or uncontrolled diseases per the Investigator's discretion
9. Evidence of GCA as indicated by typical (cranial) symptoms (e.g., persistent or recurrent localized headache, temporal artery or scalp tenderness, jaw claudication, blurry or loss of vision, symptoms of stroke), extremity claudication, imaging and/or temporal artery biopsy result

   • Note: Imaging and/or temporal artery biopsy are not standard of care for PMR management and diagnosis and are therefore not mandated as part of the screening; Patients with PMR symptoms only who have a temporal artery biopsy in line with GCA and/or radiologic signs of vasculitis may be eligible for the GCA cohort
10. Concurrent rheumatoid arthritis or other inflammatory arthritis or other connective tissue diseases, such as but not limited to systemic lupus erythematosus, systemic sclerosis, vasculitis, myositis, mixed connective tissue disease, and ankylosing spondylitis
11. Concurrent diagnosis or history of neuropathic muscular diseases including fibromyalgia
12. Inadequately treated hypothyroidism (e.g., persistence of symptoms, lack of normalization of serum TSH despite regular hormonal replacement treatment)

Additional protocol-defined inclusion / exclusion criteria may apply.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Secukinumab: Maximum concentration at steady state (Cmax,ss) | Baseline, Week 4 and Week 8: Pre-dose and End-of Infusion (EOI); Weeks 9, 10, 11, 12, 16 and 20: Anytime
  Venous whole blood samples will be collected and analyzed for all PK evaluable participants. Maximum concentration at steady state (Cmax,ss) will be listed and summarized using descriptive statistics.
Secukinumab: Minimum concentration at steady state (Cmin,ss) | Baseline, Week 4 and Week 8: Pre-dose and End-of Infusion (EOI); Weeks 9, 10, 11, 12, 16 and 20: Anytime
  Venous whole blood samples will be collected and analyzed for all PK evaluable participants. Minimum concentration at steady state (Cmin,ss) will be listed and summarized using descriptive statistics.
Secukinumab: Area under the concentration-time curve at steady state during a dosing interval (AUCtau,ss) | Baseline, Week 4 and Week 8: Pre-dose and End-of Infusion (EOI); Weeks 9, 10, 11, 12, 16 and 20: Anytime
  Venous whole blood samples will be collected and analyzed for all PK evaluable participants. Area under the concentration-time curve at steady state during a dosing interval (AUCtau,ss) will be listed and summarized using descriptive statistics.
Secukinumab: Average concentration at steady state (Cavg,ss [=AUCtau,ss/tau]) | Baseline, Week 4 and Week 8: Pre-dose and End-of Infusion (EOI); Weeks 9, 10, 11, 12, 16 and 20: Anytime
  Venous whole blood samples will be collected and analyzed for all PK evaluable participants. Average concentration at steady state (Cavg,ss [=AUCtau,ss/tau]) will be listed and summarized using descriptive statistics.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events | Up to 12 weeks after last dose administration.
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs) and Serious Adverse Event (TESAEs), through the monitoring of relevant clinical and laboratory safety parameters.
Secukinumab: Clearance (CL) | Baseline, Week 4 and Week 8: Pre-dose and End-of Infusion (EOI); Weeks 9, 10, 11, 12, 16 and 20: Anytime
  Venous whole blood samples will be collected and analyzed for all PK evaluable participants. Clearance (CL) will be listed and summarized using descriptive statistics.
Secukinumab: Volume of distribution at steady state (Vss) | Baseline, Week 4 and Week 8: Pre-dose and End-of Infusion (EOI); Weeks 9, 10, 11, 12, 16 and 20: Anytime
  Venous whole blood samples will be collected and analyzed for all PK evaluable participants. Volume of distribution at steady state (Vss) will be listed and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (8):
  - Rheumatology Associates of South Florida, Boca Raton, Florida
  - FL Medical Clinic Orlando Health, Zephyrhills, Florida
  - Willow Rheumatology Wellness, Willowbrook, Illinois
  - Altoona Center for Clin Res, Duncansville, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Accurate Clinical Research Inc, San Antonio, Texas
  - Overlake Internal Med Associates, Bellevue, Washington
  - Rheumatology Pulmonary Clinic, Beckley, West Virginia
- Czechia (2):
  - Novartis Investigative Site, Uherské Hradiště, Uherske Hradiste
  - Novartis Investigative Site, Brno-Bohunice
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Reggio Emilia, RE
- Novartis Investigative Site, Lisbon, Portugal
- Spain (2):
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CAIN457E22101 Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18407